CLINICAL TRIAL: NCT07022301
Title: A Phase II Study Evaluating the Safety and Efficacy of Sintilimab Plus Anlotinib as Second or Further-line Therapy for ES-SCLC Who Have Progressed After Anti- PD- 1/L1 Therapy
Brief Title: Sintilimab Plus Anlotinib as Second or Further-line Therapy for ES-SCLC Who Have Progressed After Anti-PD-1/L1 Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-ethics-48
Record Dates: First submitted 2025-05-22; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Small Cell Lung Cancer Extensive Stage; Resistance to Immunotherapy
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Drug: Sintilimab combined with anlotinib
  Interventions: Drug: sintilimab combined with anlotinib

INTERVENTIONS:
Drug: sintilimab combined with anlotinib — Patients who met the inclusion criteria were treated with Sintilimab plus anlotinib every 3 weeks until disease progression or intolerable adverse reactions or death(up to 24 months).

SUMMARY:
The phase II study enrolled ES-SCLC patients who had disease progression after anti-PD-1/L1 therapy. Participants received intravenous sintilimab 200 mg on day one and oral daily anlotinib 8-12 mg on days 1-14 once every three weeks per cycle. The primary endpoint was objective response rate (ORR). The secondary endpoints included overall survival (OS), progression-free survival (PFS) , disease control rate (DCR) and safety.

ELIGIBILITY:
Inclusion Criteria:

* 1. At the time of signing the informed consent form, both men and women must be at least 18 years old.
* 2. Widespread recurrent small cell lung cancer diagnosed by histology or cytology and progressing after 3 months of standard immunization.
* 3. According to RECIST 1.1 criteria, patients must have at least one measurable lesion (lesions that have undergone radiotherapy must show clear progression in order to be considered measurable lesions).
* 4. ECOG PS score: 0-1 points.
* 5. Expected survival period ≥ 3 months.
* 6. Important organ functions must meet the following standards:

  1) Blood routine examination: (No blood transfusion or use of cytokine drugs such as G-CSF for corrective treatment within 2 weeks before screening)
  1. Hemoglobin (HB) ≥ 90 g/L;
  2. Absolute neutrophil count (ANC) ≥ 1.5 × 10*9/L;
  3. Platelet count (PLT) ≥ 90 × 10*9/L;
  4. White blood cell count (WBC) ≥ 3.0 × 109/L and<15 × 10*9/L; 2) Other tests: (did not receive human serum albumin injection within 14 days before screening)
  5. AST and ALT ≤ 3 x ULN;
  6. ALP ≤ 2.5 x ULN (≤ 5 x ULN if there is bone metastasis);
  7. TBiL≤1x ULN；
  8. ALB≥30g/L；
  9. Cr ≤ 1.5 x ULN, while creatinine clearance rate (CrCL) ≥ 60mL/min (Cockcroft Gault formula);
  10. TSH ≤ 1 x ULN (if abnormal, FT3 and FT4 levels should be examined simultaneously. If FT3 and FT4 levels are normal, they can be included in the group)
  11. APTT ≤ 1.5 x ULN, while INR or PT ≤ 1.5 x ULN (not receiving anticoagulant therapy).
  12. Male QTc<450 ms, female QTc<470 ms, LVEF ≥ 50%
* 7. Non surgical sterilization or female patients of childbearing age must undergo a serum pregnancy test within 3 days before the first medication, and the result must be negative; And it must be non lactating. Female patients of childbearing age or male patients with partners of childbearing age must agree to use efficient contraception methods during the study period and within 6 months after the last administration of the study drug.
* 8. The patient voluntarily joined this clinical study and signed an informed consent form, with good compliance and the ability to cooperate with follow-up.

Exclusion Criteria:

* 1. Imaging shows that the tumor has invaded large blood vessels or has unclear boundaries with blood vessels.
* 2. Imaging shows the presence of obvious pulmonary hollow or necrotic tumors.
* 3. Symptomatic central nervous system metastases (such as brain metastases or meningeal metastases).
* 4. Patients with conditions such as malignant meningitis and spinal cord compression.
* 5. Persons who have suffered from other malignant tumors in the past or at the same time, unless they are skin basal cell carcinoma, superficial bladder cancer, skin squamous cell carcinoma, cervical carcinoma in situ or other carcinoma in situ that have achieved complete remission at least 5 years before screening and do not need or are not expected to need other treatment during the study period.
* 6. Those who have had or currently have objective evidence of idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, tissue pneumonitis (such as bronchitis, occlusive vasculitis), drug-induced pneumonia, or screening period CT showing active pneumonia or lung function examination confirming severe impairment of lung function.
* 7. Individuals with any active, known or suspected autoimmune diseases (including but not limited to: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, enteritis, multiple sclerosis, vasculitis, glomerulonephritis, uveitis, pituitary inflammation, hyperthyroidism, etc.). Type I diabetes patients who are allowed to receive stabilizing dose insulin treatment, hypothyroidism patients who only need hormone replacement treatment, and skin diseases (such as eczema, vitiligo, or psoriasis) that do not require systemic treatment and have no acute deterioration within 1 year before the screening period.
* 8. Patients suspected of having active pulmonary tuberculosis should undergo chest X-ray, sputum examination, and exclusion based on clinical symptoms and signs. Individuals with a history of active pulmonary tuberculosis infection within the previous year should be excluded, even if they have been treated; Subjects with a history of active pulmonary tuberculosis infection more than one year ago should also be excluded unless it is proven that the previous course and type of anti tuberculosis treatment used were appropriate.
* 9. Clinical symptoms or diseases of the heart that have not been well controlled, such as: (1) NYHA grade 2 or above heart failure, (2) unstable angina, (3) myocardial infarction within 1 year, and (4) clinically significant supraventricular or ventricular arrhythmias that require treatment or intervention.
* 10. Patients with hypertension who cannot achieve good control with antihypertensive medication (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg).
* 11. Urine routine showed urinary protein ≥++, and 24-hour urinary protein quantification was confirmed to be>1.0 g through quantitative detection of urinary protein.
* 12. For individuals with a tendency towards thrombosis or undergoing thrombolytic/anticoagulant therapy, prophylactic use of low-dose aspirin (≤ 100mg/d) and low molecular weight heparin (≤ 40mg/d) is allowed.
* 13. Those who have received>30 Gy of chest radiation therapy within the first 6 months of randomization, and have undergone major surgical treatment within the first 4 weeks of randomization, but have not recovered from the toxicity and/or complications of previous intervention measures to NCI-CTC AE ≤ 1 degree (except for hair loss and indicators clearly defined in the inclusion criteria).
* 14. Within the first 6 months of randomization, there have been arterial/venous thrombotic events, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism.
* 15. Individuals with a daily cough/hemoptysis volume greater than 2.5mL within the first month of randomization. Individuals with a history of hereditary or acquired bleeding or coagulation dysfunction. Within the first 3 months of randomization, there have been significant clinical bleeding symptoms or clear bleeding tendencies, such as gastrointestinal bleeding, hemorrhagic gastric ulcers, etc.
* 16. Participants who have experienced severe infections within the previous month prior to randomization, including but not limited to infection complications requiring hospitalization, bacteremia, severe pneumonia, etc; Subjects with any active infection, or experiencing unexplained fever>38.5 ℃ during screening or before the first dose.
* 17. Patients who have received anti-tumor vaccines or other immunomodulatory drugs (such as interleukin-2, thymosin, shiitake polysaccharides, etc.) within the previous month of randomization, or patients who will receive attenuated live vaccines.
* 18. Subjects who have received systemic therapy with corticosteroids (>10 mg/day of prednisone or other equivalent hormones) or other immunosuppressive agents within the previous month prior to randomization. In the absence of active autoimmune diseases, inhalation or topical use of corticosteroids, as well as adrenal hormone replacement therapy with a dose ≤ 10 mg/day of prednisone efficacy dose, are allowed.
* 19. Known to have a positive history of human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS). It is known that there is active hepatitis or co infection with hepatitis B and hepatitis C. (hepatitis B reference: HBsAg is positive, and the HBV DNA detection value exceeds the upper limit of normal value; Hepatitis C reference: HCV antibody positive and HCV virus titer detection value exceeding the upper limit of normal.
* 20. are known to have experienced allergic reactions to other monoclonal antibodies or any component of anlotinib.
* 21. Those who are currently participating in other clinical studies or have been randomized for less than 4 weeks (or 5 half lives of the study drug) since the end of the previous clinical study (last dose);
* 22. According to the researchers' assessment, there are other factors that may affect the research results or lead to the forced termination of this study, such as alcohol abuse, drug use, drug abuse, other serious illnesses (including mental illnesses) that require concurrent treatment, serious laboratory test abnormalities, and family or social factors that may affect medication safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 months
  the rate of patients with PR and CR

SECONDARY OUTCOMES:
OS | 24 months
  The time from the beginning of treatment to the time when the patient dies from any cause
PFS | 24 months
  The time from the beginning of treatment to the time when the disease progresses or the patient dies from any cause
AE | 24 months
  Safety will be evaluated by AE

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38516099/